CLINICAL TRIAL: NCT00297973
Title: Cardiovascular Risk Assessment In Patients With Hypertension And At Least Three Other Risk Factors, Treated With Caduet Compared To Usual Care: The Right Study
Brief Title: Cardiovascular Risk Assessment in Patients Treated With Caduet
Acronym: RIGHT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: A3841038
Record Dates: First submitted 2006-02-27; First posted 2006-03-01 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Blood Pressure; Blood Specimen Collection

INTERVENTIONS:
Procedure: Blood pressure measurements
Procedure: Blood samples

SUMMARY:
Compare the reduction in Framingham's predicted 10-year risk of a coronary event (6) in patients with hypertension and at least three other cardiovascular risk factors (including diabetic patients) seen in private practice and randomized to either Caduet or usual care.

ELIGIBILITY:
Inclusion Criteria:

* 1.Male or female, 18 years of age or over, 2.Patient with hypertension and at least three other CV risk factors, 3.Hypertension, treated or not, but not at the currently recommended goals (140/90 mmHg for most patients, 130/80 mmHg for patients with diabetes or nephropathy). In case of treated hypertension, patients should be on their current treatment for at least 4 weeks before randomisation,

Exclusion Criteria:

* 1. Patient with a history of coronary heart disease, 2.Patients with a history of familial hypercholesterolemia, 3.Patient with malignant HTN, 4.Non-essential hypertension, 5.Known hypersensitivity to dihydropyridines, 6.Patients already receiving a dihydropyridine, 7.Known hypersensitivity to HMG-CoA-reductase inhibitors, 8.Patients currently receiving or who has received a HMG-CoA-reductase within the 3 months prior to selection, 9.Patients currently receiving or who has received a fibric acid, resins, ezetimibe, nicotinic acid and all other drug which is known to affect lipid levels, within 6 weeks prior to selection,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1442 (Actual)
Dates: Start 2006-02; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
% reduction in Framingham's predicted 10-year risk of a coronary event between V1 and V3 in the Caduet group compared to the usual care group (6) (including diabetic patients)

SECONDARY OUTCOMES:
1. % patients changing risk category between V1 and V3 2. % reduction in Framingham's predicted 10-year risk of a coronary event (8) excluding diabetic patients 3. Clinical and biological safety during treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (342):
- France (342):
  - Pfizer Investigational Site, Abbeville
  - Pfizer Investigational Site, Aire-sur-la-Lys
  - Pfizer Investigational Site, Aix-les-Bains
  - Pfizer Investigational Site, Alençon
  - Pfizer Investigational Site, Allaire
  - Pfizer Investigational Site, Amboise
  - Pfizer Investigational Site, Amiens
  - Pfizer Investigational Site, Andrézieux-Bouthéon
  - Pfizer Investigational Site, Angers
  - Pfizer Investigational Site, Annecy
  - Pfizer Investigational Site, Annecy-le-Vieux
  - Pfizer Investigational Site, Annemasse
  - Pfizer Investigational Site, Anzin
  - Pfizer Investigational Site, Appoigny
  - Pfizer Investigational Site, Apt
  - Pfizer Investigational Site, Argenteuil
  - Pfizer Investigational Site, Arles
  - Pfizer Investigational Site, Arnèke
  - Pfizer Investigational Site, Arpajon
  - Pfizer Investigational Site, Arsac
  - Pfizer Investigational Site, Aubagne
  - Pfizer Investigational Site, Auchel
  - Pfizer Investigational Site, Audresselles
  - Pfizer Investigational Site, Autrans
  - Pfizer Investigational Site, Balma
  - Pfizer Investigational Site, Bastia
  - Pfizer Investigational Site, Bayonne
  - Pfizer Investigational Site, Beaucaire
  - Pfizer Investigational Site, Beaumont-lès-Valence
  - Pfizer Investigational Site, Beaurains
  - Pfizer Investigational Site, Beausoleil
  - Pfizer Investigational Site, Belley
  - Pfizer Investigational Site, Belpech
  - Pfizer Investigational Site, Benquet
  - Pfizer Investigational Site, Berck
  - Pfizer Investigational Site, Bersée
  - Pfizer Investigational Site, Béthune
  - Pfizer Investigational Site, Béziers
  - Pfizer Investigational Site, Biarritz
  - Pfizer Investigational Site, Blasimon
  - Pfizer Investigational Site, Blois
  - Pfizer Investigational Site, Boën-sur-Lignon
  - Pfizer Investigational Site, Bondues
  - Pfizer Investigational Site, Bondy
  - Pfizer Investigational Site, Bordeaux
  - Pfizer Investigational Site, Bourg-Saint-Andéol
  - Pfizer Investigational Site, Bourges
  - Pfizer Investigational Site, Brest
  - Pfizer Investigational Site, Bréhan
  - Pfizer Investigational Site, Brignoud
  - Pfizer Investigational Site, Bruay-la-Buissière
  - Pfizer Investigational Site, Bœrsch
  - Pfizer Investigational Site, Cabestany
  - Pfizer Investigational Site, Caen
  - Pfizer Investigational Site, Cagnes-sur-Mer
  - Pfizer Investigational Site, Cannes
  - Pfizer Investigational Site, Cannes La Bocca
  - Pfizer Investigational Site, Carnon-Plage
  - Pfizer Investigational Site, Castelnau Le Fez
  - Pfizer Investigational Site, Castelsarrasin
  - Pfizer Investigational Site, Castres
  - Pfizer Investigational Site, Caylus
  - Pfizer Investigational Site, Cergy
  - Pfizer Investigational Site, Cestas
  - Pfizer Investigational Site, Champagne-au-Mont-d'Or
  - Pfizer Investigational Site, Chanceaux-sur-Choisille
  - Pfizer Investigational Site, Charleville-Mézières
  - Pfizer Investigational Site, Chartres
  - Pfizer Investigational Site, Chatou
  - Pfizer Investigational Site, Chelles
  - Pfizer Investigational Site, Chenôve
  - Pfizer Investigational Site, Chilly-Mazarin
  - Pfizer Investigational Site, Clairac
  - Pfizer Investigational Site, Clary
  - Pfizer Investigational Site, Clermont-Ferrand
  - Pfizer Investigational Site, Collioure
  - Pfizer Investigational Site, Colombier-Fontaine
  - Pfizer Investigational Site, Colomiers
  - Pfizer Investigational Site, Condat-sur-Vienne
  - Pfizer Investigational Site, Courthézon
  - Pfizer Investigational Site, Craponne
  - Pfizer Investigational Site, Crest
  - Pfizer Investigational Site, Crécy-la-Chapelle
  - Pfizer Investigational Site, Créteil
  - Pfizer Investigational Site, Crotenay
  - Pfizer Investigational Site, Cuise-la-Motte
  - Pfizer Investigational Site, Denain
  - Pfizer Investigational Site, Dijon
  - Pfizer Investigational Site, Dugny-sur-Meuse
  - Pfizer Investigational Site, Dunkirk
  - Pfizer Investigational Site, Eckbolsheim
  - Pfizer Investigational Site, Eckwersheim
  - Pfizer Investigational Site, Échirolles
  - Pfizer Investigational Site, Épernay
  - Pfizer Investigational Site, Épinal
  - Pfizer Investigational Site, Épinay-sur-Seine
  - Pfizer Investigational Site, Étampes
  - Pfizer Investigational Site, Étang-sur-Arroux
  - Pfizer Investigational Site, Évreux
  - Pfizer Investigational Site, Falaise
  - Pfizer Investigational Site, Fayence
  - Pfizer Investigational Site, Fenioux
  - Pfizer Investigational Site, Ferney-Voltaire
  - Pfizer Investigational Site, Floirac
  - Pfizer Investigational Site, Fontaine
  - Pfizer Investigational Site, Fontaine-lès-Dijon
  - Pfizer Investigational Site, Fontainebleau
  - Pfizer Investigational Site, Fontenay-sous-Bois
  - Pfizer Investigational Site, Fontès
  - Pfizer Investigational Site, Fos-sur-Mer
  - Pfizer Investigational Site, Franconville
  - Pfizer Investigational Site, Fumay
  - Pfizer Investigational Site, Gaillefontaine
  - Pfizer Investigational Site, Gambsheim
  - Pfizer Investigational Site, Gap
  - Pfizer Investigational Site, Gonesse
  - Pfizer Investigational Site, Gonneville-la-Mallet
  - Pfizer Investigational Site, Gradignan
  - Pfizer Investigational Site, Grand-Couronne
  - Pfizer Investigational Site, Grendelbruch
  - Pfizer Investigational Site, Grenoble
  - Pfizer Investigational Site, Gréasque
  - Pfizer Investigational Site, Groslay
  - Pfizer Investigational Site, Guise
  - Pfizer Investigational Site, Haguenau
  - Pfizer Investigational Site, Harnes
  - Pfizer Investigational Site, Hasparren
  - Pfizer Investigational Site, Hautmont
  - Pfizer Investigational Site, Hochfelden
  - Pfizer Investigational Site, Hostens
  - Pfizer Investigational Site, Ivry-sur-Seine
  - Pfizer Investigational Site, Jargeau
  - Pfizer Investigational Site, Jarville-la-Malgrange
  - Pfizer Investigational Site, Jeumont
  - Pfizer Investigational Site, L'Isle-sur-la-Sorgue
  - Pfizer Investigational Site, La Baule-Escoublac
  - Pfizer Investigational Site, La Chapelle-des-Marais
  - Pfizer Investigational Site, La Chapelle-sur-Erdre
  - Pfizer Investigational Site, La Ciotat
  - Pfizer Investigational Site, La Courneuve
  - Pfizer Investigational Site, La Crèche
  - Pfizer Investigational Site, La Fère
  - Pfizer Investigational Site, La Francheville
  - Pfizer Investigational Site, La Grande-Motte
  - Pfizer Investigational Site, La Grande-Paroisse
  - Pfizer Investigational Site, La Rochelle
  - Pfizer Investigational Site, La Tour-du-Crieu
  - Pfizer Investigational Site, La Trinité-sur-Mer
  - Pfizer Investigational Site, Labastidette
  - Pfizer Investigational Site, Lacrouzette
  - Pfizer Investigational Site, Lamagistère
  - Pfizer Investigational Site, Lamarque
  - Pfizer Investigational Site, Langon
  - Pfizer Investigational Site, Lattes
  - Pfizer Investigational Site, Laval
  - Pfizer Investigational Site, Lavernose-Lacasse
  - Pfizer Investigational Site, Laxou
  - Pfizer Investigational Site, Le Bourget
  - Pfizer Investigational Site, Le Cannet
  - Pfizer Investigational Site, Le Havre
  - Pfizer Investigational Site, Lembeye
  - Pfizer Investigational Site, Les Issambres
  - Pfizer Investigational Site, Les Sables-d'Olonne
  - Pfizer Investigational Site, Lesquin
  - Pfizer Investigational Site, Liancourt
  - Pfizer Investigational Site, Ligny-en-Barrois
  - Pfizer Investigational Site, Lille
  - Pfizer Investigational Site, Limoges
  - Pfizer Investigational Site, Lorient
  - Pfizer Investigational Site, Lourdes
  - Pfizer Investigational Site, Lucheux
  - Pfizer Investigational Site, Luxeuil-les-Bains
  - Pfizer Investigational Site, Lyon
  - Pfizer Investigational Site, Mandelieu-la-Napoule
  - Pfizer Investigational Site, Marcq-en-Barœul
  - Pfizer Investigational Site, Marseille
  - Pfizer Investigational Site, Martigues
  - Pfizer Investigational Site, Masseret
  - Pfizer Investigational Site, Mauguio
  - Pfizer Investigational Site, Meaux Beauval
  - Pfizer Investigational Site, Meaux-Beauval
  - Pfizer Investigational Site, Mennecy
  - Pfizer Investigational Site, Mensignac
  - Pfizer Investigational Site, Merlimont
  - Pfizer Investigational Site, Metz
  - Pfizer Investigational Site, Mirabel-et-Blacons
  - Pfizer Investigational Site, Miramas
  - Pfizer Investigational Site, Miramont-de-Guyenne
  - Pfizer Investigational Site, Mittersheim
  - Pfizer Investigational Site, Mommenheim
  - Pfizer Investigational Site, Mons-en-Barœul
  - Pfizer Investigational Site, Montauroux
  - Pfizer Investigational Site, Montbéliard
  - Pfizer Investigational Site, Monteux
  - Pfizer Investigational Site, Montpellier
  - Pfizer Investigational Site, Montreuil
  - Pfizer Investigational Site, Montrevel-en-Bresse
  - Pfizer Investigational Site, Moreuil
  - Pfizer Investigational Site, Morlaix
  - Pfizer Investigational Site, Mourenx
  - Pfizer Investigational Site, Muespach
  - Pfizer Investigational Site, Mulhouse
  - Pfizer Investigational Site, Mundolsheim
  - Pfizer Investigational Site, Nancy
  - Pfizer Investigational Site, Nantes
  - Pfizer Investigational Site, Nevers
  - Pfizer Investigational Site, Néris-les-Bains
  - Pfizer Investigational Site, Nice
  - Pfizer Investigational Site, Niort
  - Pfizer Investigational Site, Nogent-sur-Marne
  - Pfizer Investigational Site, Noisiel
  - Pfizer Investigational Site, Noyon
  - Pfizer Investigational Site, Oberhausbergen
  - Pfizer Investigational Site, Obernai
  - Pfizer Investigational Site, Objat
  - Pfizer Investigational Site, Orange
  - Pfizer Investigational Site, Orchamps
  - Pfizer Investigational Site, Orry-la-Ville
  - Pfizer Investigational Site, Ossès
  - Pfizer Investigational Site, Pacy-sur-Eure
  - Pfizer Investigational Site, Palau-del-Vidre
  - Pfizer Investigational Site, Paris
  - Pfizer Investigational Site, Parthenay
  - Pfizer Investigational Site, Perpignan
  - Pfizer Investigational Site, Pessac
  - Pfizer Investigational Site, Petit-Couronne
  - Pfizer Investigational Site, Pfulgriesheim
  - Pfizer Investigational Site, Phalempin
  - Pfizer Investigational Site, Pont-à-Mousson
  - Pfizer Investigational Site, Portet-sur-Garonne
  - Pfizer Investigational Site, Porto-Vecchio
  - Pfizer Investigational Site, Poussan
  - Pfizer Investigational Site, Pradines
  - Pfizer Investigational Site, Précy-sur-Oise
  - Pfizer Investigational Site, Quimperlé
  - Pfizer Investigational Site, Rebais
  - Pfizer Investigational Site, Reims
  - Pfizer Investigational Site, Remiremont
  - Pfizer Investigational Site, Rennes
  - Pfizer Investigational Site, Rigney
  - Pfizer Investigational Site, Rodez
  - Pfizer Investigational Site, Rognac
  - Pfizer Investigational Site, Rohrwiller
  - Pfizer Investigational Site, Romans-sur-Isère
  - Pfizer Investigational Site, Roncq
  - Pfizer Investigational Site, Roquevaire
  - Pfizer Investigational Site, Roubaix
  - Pfizer Investigational Site, Rozay-en-Brie
  - Pfizer Investigational Site, Saint-Agrève
  - Pfizer Investigational Site, Saint-Avold
  - Pfizer Investigational Site, Saint-Brieuc
  - Pfizer Investigational Site, Saint-Denis
  - Pfizer Investigational Site, Saint-Dié
  - Pfizer Investigational Site, Saint-Erme-Outre-et-Ramecourt
  - Pfizer Investigational Site, Saint-Etienne
  - Pfizer Investigational Site, Saint-Fons
  - Pfizer Investigational Site, Saint-Germain-au-Mont-d'Or
  - Pfizer Investigational Site, Saint-Germain-de-Marencennes
  - Pfizer Investigational Site, Saint-Girons
  - Pfizer Investigational Site, Saint-Jean-de-Braye
  - Pfizer Investigational Site, Saint-Jean-de-Luz
  - Pfizer Investigational Site, Saint-Jean-de-Maurienne
  - Pfizer Investigational Site, Saint-Joachim
  - Pfizer Investigational Site, Saint-Leu-d'Esserent
  - Pfizer Investigational Site, Saint-Leu-la-Forêt
  - Pfizer Investigational Site, Saint-Marcel-lès-Valence
  - Pfizer Investigational Site, Saint-Martin-d'Hères
  - Pfizer Investigational Site, Saint-Martin-d'Oney
  - Pfizer Investigational Site, Saint-Martin-des-Champs
  - Pfizer Investigational Site, Saint-Martin-du-Bois
  - Pfizer Investigational Site, Saint-Morillon
  - Pfizer Investigational Site, Saint-Ouen
  - Pfizer Investigational Site, Saint-Ouen-l'Aumône
  - Pfizer Investigational Site, Saint-Rambert-d'Albon
  - Pfizer Investigational Site, Saint-Raphaël
  - Pfizer Investigational Site, Saint-Rémy-de-Provence
  - Pfizer Investigational Site, Saint-Saulve
  - Pfizer Investigational Site, Saint-Sébastien-sur-Loire
  - Pfizer Investigational Site, Saint-Sulpice-la-Pointe
  - Pfizer Investigational Site, Saint-Tropez
  - Pfizer Investigational Site, Saint-Yrieix-la-Perche
  - Pfizer Investigational Site, Salles
  - Pfizer Investigational Site, Salon-de-Provence
  - Pfizer Investigational Site, Sanary-sur-Mer
  - Pfizer Investigational Site, Sarlat-la-Canéda
  - Pfizer Investigational Site, Sartrouville
  - Pfizer Investigational Site, Schweighouse-sur-Moder
  - Pfizer Investigational Site, Semur-en-Auxois
  - Pfizer Investigational Site, Sevrier
  - Pfizer Investigational Site, Sète
  - Pfizer Investigational Site, Sélestat
  - Pfizer Investigational Site, Soissons
  - Pfizer Investigational Site, Solgne
  - Pfizer Investigational Site, Ste. Maxime
  - Pfizer Investigational Site, Ste. Suzanne
  - Pfizer Investigational Site, Strasbourg
  - Pfizer Investigational Site, Suresnes
  - Pfizer Investigational Site, Targon
  - Pfizer Investigational Site, Tergnier
  - Pfizer Investigational Site, Thiant
  - Pfizer Investigational Site, Thierville-sur-Meuse
  - Pfizer Investigational Site, Thiviers
  - Pfizer Investigational Site, Thônes
  - Pfizer Investigational Site, Toul
  - Pfizer Investigational Site, Toulon
  - Pfizer Investigational Site, Toulouse
  - Pfizer Investigational Site, Tours
  - Pfizer Investigational Site, Trie-sur-Baïse
  - Pfizer Investigational Site, Vabres-l'Abbaye
  - Pfizer Investigational Site, Vacqueyras
  - Pfizer Investigational Site, Vagney
  - Pfizer Investigational Site, Valenciennes
  - Pfizer Investigational Site, Valognes
  - Pfizer Investigational Site, Valréas
  - Pfizer Investigational Site, Vals-les-Bains
  - Pfizer Investigational Site, Vandœuvre-lès-Nancy
  - Pfizer Investigational Site, Vannes
  - Pfizer Investigational Site, Varces-Allières-et-Risset
  - Pfizer Investigational Site, Vatan
  - Pfizer Investigational Site, Vence
  - Pfizer Investigational Site, Vernet
  - Pfizer Investigational Site, Vélines
  - Pfizer Investigational Site, Vélizy-Villacoublay
  - Pfizer Investigational Site, Vénissieux
  - Pfizer Investigational Site, Viane
  - Pfizer Investigational Site, Villard-Bonnot
  - Pfizer Investigational Site, Villefranche-de-Rouergue
  - Pfizer Investigational Site, Villefranche-sur-Mer
  - Pfizer Investigational Site, Villefranche-sur-Saône
  - Pfizer Investigational Site, Villeneuve-lès-Maguelone
  - Pfizer Investigational Site, Villeparisis
  - Pfizer Investigational Site, Villers-Saint-Paul
  - Pfizer Investigational Site, Villette-d'Anthon
  - Pfizer Investigational Site, Viry-Châtillon
  - Pfizer Investigational Site, Vitrolles
  - Pfizer Investigational Site, Vix
  - Pfizer Investigational Site, Wambrechies
  - Pfizer Investigational Site, Wasselonne
  - Pfizer Investigational Site, Wattignies
  - Pfizer Investigational Site, Wattrelos
  - Pfizer Investigational Site, Witry-lès-Reims
  - Pfizer Investigational Site, Yffiniac

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3841038&StudyName=Cardiovascular%20Risk%20Assessment%20in%20patients%20treated%20with%20Caduet